CLINICAL TRIAL: NCT00455468
Title: Randomized Controlled Trial (RCT) in Children With Severe Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Principal Investigator, International Centre for Diarrhoeal Disease Research, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-037
Record Dates: First submitted 2007-04-01; First posted 2007-04-03 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2007-03

CONDITIONS: Severe Pneumonia
Keywords: Severe pneumonia; children; day care management; hospitalized management; Randomized controlled trial; Under five children
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Day-care treatment vs. hospital care

SUMMARY:
Pneumonia is the leading cause of childhood morbidity and death in many developing countries including Bangladesh, causing about 2 million deaths worldwide each year. Pneumonia is an infection of the lungs, most commonly caused by viruses or bacteria like Streptococcus pneumoniae and Haemophilus influenzae. Depending on the clinical presentation, pneumonia can be classified as very severe, severe or non-severe, with specific treatment for each of them except for antibiotic therapy. Severe and very severe pneumonia require hospitalization for additional supportive treatment such as suction, oxygen therapy and administration of bronchodilator. In Bangladesh, the number of hospital beds is inadequate for admission of all pneumonia cases that require hospitalization; however, it is also important to provide institutional care to those children who cannot be hospitalized due to bed constraints. Provision of appropriate antibiotics and supportive cares during the period of stay at established day-care centres could be an effective alternative. The impetus for this study came from the findings of our recently completed study titled "Daycare-based management of severe pneumonia in under-5 children when hospitalization is not possible due to the lack of beds". This study successfully managed children (n=251), but it was not a randomized trial and thus direct comparison of the efficacy of management of severe pneumonia at the day-care centre, essential for building confidence for implementing this management policy, is not possible. We, the researchers at the International Centre for Diarrhoeal Disease Research, Bangladesh, could not plan a randomized, controlled trial (RCT) because of ethical reasons. Now that we have data suggesting effectiveness as well as safety of the day-care based treatment for management of children with severe pneumonia, a RCT should be possible. Two hundred fifty-one children with severe pneumonia were enrolled at the Radda Clinic from June 2003 to May 2005. The mean age was 7±7 (2-55) months, 86% infants, 63% boys and 91% breast-fed. History of cough was present in 99% cases, fever in 89% and rapid breathing in 67% cases. Forty-four percent of children were febrile (≥38°C), 93% children had vesicular breath sound and 99% bilateral rales. Fifty-seven percent of children were hypoxic with mean oxygen saturation of (93±4)%, which was corrected by oxygen therapy (98±3)%. Eighty percent of children had severe pneumonia and 20% had very severe pneumonia. The mean duration of clinic stay was (7±2) days. Two hundred thirty-four (93%) children completed the study successfully, 11 (4.4%) referred to hospitals (only one participant had to visit hospital at night due to deterioration of his condition, 9 were referred to hospital at the time of clinic closure i.e., at 5 pm and one participant was referred to hospital during the morning hours) and 6 (2.4%) left against medical advice (LAMA). There was no death during the period of clinic stay but only four (1.6%) deaths occurred during the 3 months follow-up. The study indicated that treatment of severe pneumonia in children at the day-care centre is effective and safe and thus it is comparable to the hospital care. If the day-care based management is found to have comparable efficacy to that of hospitalized management of severe pneumonia in children then they could be managed at outpatient, day-care set ups reducing hospitalization and thus freeing beds for management of other children who need hospitalized care. Additionally, availability of the treatment facility in community set-ups will be cost and time saving for the population. Children of either sex, aged 2-59 months, attending the Radda Clinic and Institute of Child Health and Shishu Hospital (ICHSH) with severe pneumonia will be randomized to receive either the day-care management at the clinic or hospitalized management at the ICHSH. Children randomized to receive day-care treatment will stay at the clinic from 8 am-5 pm and will receive antibiotics and other supportive cares. At 5 pm, they would be send to respective homes with advice to bring back their children to the clinic next morning, and advised to provide other supports at home. The same management would be continued till improvement and discharged and followed up every 2 weeks for 3 months. Children randomized to receive hospitalized management would be admitted at ICHSH and receive standard treatment like antibiotics and other supportive cares. The same treatment would be continued for 24 hours/day (rather than 9 hours/day at the day-care clinic) till improvement and discharged and followed-up at the ICHSH every 2 weeks for 3 months. About 3000 children with pneumonia visit Radda Clinic each year and about 200 of them will have severe pneumonia requiring hospitalization. Thus, we hope to enroll 368 (184 in each site) children with severe pneumonia during a 2-year study period.

DETAILED DESCRIPTION:
Acute lower respiratory infection (ALRI), particularly pneumonia is the leading cause of childhood morbidity and death in the developing countries including Bangladesh. Acute respiratory infection (ARI) causes more than 2 million child deaths worldwide each year; most of these deaths are due to pneumonia and 90% of them occur in less-developed countries. Recent estimates suggest that 1.9 million (95% CI 1.6-2.2 million) children died from ARI throughout the world in 2000, and 70% of them occurred in Africa and Southeast Asia. ARI is also a major cause of visits to the outpatient and emergency departments as well as admissions to the hospitals. Although bronchiolitis, tracheobronchitis and pneumonia, each accounts for about one-third of ALRI cases, pneumonia is responsible for most ALRI deaths. Three studies that reported diagnoses in children who died of ALRI revealed that a median of 89% (range 71% to 100%) of ALRI deaths were associated with pneumonia. In Bangladesh, ALRI accounts for 25% of under-5 children deaths and 40% of infantile deaths. In a study conducted at the Dhaka Hospital of the International Centre for Diarrhoeal Disease Research, Bangladesh (ICDDR,B) in 1986-88 among 401 under-5 children with ALRI, it has been observed that the most common manifestation was pneumonia and a respiratory pathogen (both bacterial and viral) was identified in 30% cases. The case fatality rates were 14% in bacterial pneumonia and 3% in viral pneumonia. Bacterial infections play a major role as a cause of pneumonia in children in developing countries. Pooled data from lung aspiration studies, mostly from developing countries, reported 52-62% isolation rates of bacteria. The case-fatality rate in severe ALRI in children aged 1-4 years is 10-15 times higher in the developing than in the developed countries. It is an infection of the lungs, most commonly caused by viruses or bacteria. It is usually not possible to determine the specific cause of pneumonia by either clinical or chest X-ray features. In children, Streptococcus pneumoniae and Haemophilus influenzae are the two most important bacterial pathogens. Respiratory Syncytial Virus (RSV) is also an important cause of ARI among preschool children. Emerging evidence suggests that Mycoplasma pneumoniae and Chlamydia pneumoniae may cause pneumonia among older children. Available data also suggests that mixed viral and bacterial infections are common in children in developing countries, which need to be treated with antibiotics. More recently, data from a large vaccine trial suggested Streptococcus pneumoniae to play a major role in the development of pneumonia associated with viral infections. The WHO recommendations for treatment of pneumonia are based on data that Streptococcus pneumoniae and Haemophilus influenzae are the most common causes of bacterial pneumonia in developing countries. Depending on clinical presentation, pneumonia can be classified as very severe, severe or non-severe with specific treatment guidelines available for each of them. The WHO defines very severe pneumonia as clinical symptoms and signs of pneumonia (cough or difficulty breathing with one or more danger signs like cyanosis, convulsions, drowsiness, stridor in calm child or inability to drink, all signifying hypoxaemia or severe respiratory distress) and severe clinical malnutrition. Severe pneumonia is defined as cough or difficulty breathing with lower chest wall in drawing with or without fast breathing defined as the respiratory rate ≥ 50 breaths per minute for children aged 2-11 months and ≥ 40 breaths per minute for children aged 12-59 months. Lower chest wall in drawing is defined as inward movement of the bony structures of the lower chest wall with inspiration, observed while the child is at rest. Finally, non-severe pneumonia is defined as cough or difficulty breathing with fast breathing as defined earlier. Antibiotic therapy is indicated irrespective of the severity of pneumonia. Proper management of children presenting in health centres and hospitals with respiratory symptoms is the cornerstone of acute respiratory infection control. To address the high mortality associated with ALRI, WHO launched a programme for control of ARI with the major objective to reduce the child mortality and to promote rational use of antibiotic. Current standard ARI case management recommends that children with cough and normal breathing be treated as outpatients without any antibiotics assuming viral infection or mild bacterial infections; those with rapid respiration (tachypnoea) indicating lower respiratory infection or pneumonia be treated with an antibiotic on an ambulatory basis (non-severe pneumonia); while those with chest wall in drawing (indicative of severe pneumonia) be admitted to hospital and treated with parenteral antibiotics and supportive cares. Vaccination against measles, pertussis, Haemophilus influenzae type b (Hib) and Streptococcus pneumoniae can help decrease the incidence and lessen the severity of respiratory infections. However, newer vaccines against respiratory infections such as Hib and pneumococcal conjugate vaccines are not widely available in developing countries. Under-5 children with respiratory symptoms are brought to the general practitioners as well as to primary health care facilities for treatment. At these respective places, the health care providers are required to differentiate between acute upper respiratory infections (AURI) and acute lower respiratory infections (ALRI)/pneumonia, and categorize severity of pneumonia taking into consideration the nutritional status of the patients and provide either ambulatory therapy or refer patients for hospitalization, as appropriate.

Severe and very severe pneumonia require hospitalization for additional supportive treatment like oro or nasopharyngeal suction, when indicated, using a suction device; oxygen therapy to hypoxic children, bronchodilators to patients with bronchospasm, bronchodilatation by nebulizer if the patients fulfill the criteria for nebulization, and fluid and nutritional management and close monitoring. In Bangladesh, the number of hospital beds are inadequate for admission of all pneumonia cases that fulfill the criteria for hospitalization. Hospitalization may also not be possible for inability of the parents to visit a hospital due to distance or, financial reason(s), despite appropriate referral. However, it is also important to provide institutional care to those children who cannot be hospitalized, at least until stabilization of their acute conditions. If such children are sent home with antibiotics, it would be important to establish an expensive, home follow up system, without which a significant proportion of them would be expected to have a fatal outcome. Provision of broad-spectrum antibiotics and appropriate supportive care during the period of stay at established day-care centres could be an effective alternative. To examine this possibility, we have recently completed a study entitled "Daycare-based management of severe pneumonia in under-5 children when hospitalization is not possible due to the lack of beds" (ICDDR,B Protocol No. 2002-036) at the Radda MCH-FP Centre, located in Mirpur Section-10, Dhaka, Bangladesh. The estimated catchment population of the Radda Clinic is about 1.5 million. The hypothesis of our recently completed study was that it would be possible to provide effective treatment and care to under-5 children with severe pneumonia at a day-care clinic set up, and if so, the need for hospitalization could be significantly reduced. The study examined if children, who required hospitalization according to WHO guidelines but were not hospitalized due to any reason, could be managed at a day-care facility (modified primary care set up), which is important to reduce morbidity and more importantly deaths among such children. We are impressed with the results, which suggested that this model of management is effective. 251 children with severe pneumonia were enrolled at the Radda Clinic from June 2003 to May 2005. The mean age was 7±7 (2-55) months, 86% were infants, 63% boys, and 91% breast-fed. On admission, history of cough was present in 99% cases, fever in 89%, rapid breathing in 67% and difficulty in breathing in 33% cases. On examination, 44% children were febrile (≥38°C), 97% children had tachypnoea with respiratory rate ≥ 50 per minute and 98% had lower chest wall in drawing. On auscultation, 93% children had vesicular breath sound and 99% bilateral rales. Most children were well nourished but 57% were hypoxic with mean oxygen saturation of (93±4)% on admission, which was corrected by oxygen therapy (98±3)%. According to WHO criteria, 80% children had severe pneumonia and 20% had very severe pneumonia. The mean duration of clinic stay was (7±2) days. 234 (93%) children completed the study successfully without any problem, 11 (4.4%) referred to hospitals (only one participant had to visit hospital at night due to deterioration of his condition, 9 were referred to hospital at the time of clinic closure i.e., at 5 pm and one participant was referred to hospital during the morning hours), and 6 (2.4%) left against medical advice (LAMA). There was no death during the period of clinic stay but only four (1.6%) deaths occurred during the 3 months follow-up period after discharge from the clinic. This study indicated that treatment of severe pneumonia in children at the day-care centre is effective and safe and thus it is comparable to the hospital care. Although this study successfully managed all children (n=251), but it was not a randomized trial and thus direct comparison of the effectiveness of management of severe pneumonia at the day-care centre, essential to recommend implementation of this management policy, is not possible. We could not plan for a RCT due to ethical reasons for our recently completed day-care pneumonia study. Now that we have data suggesting effectiveness as well as safety of the day-care based treatment and care of under-5 children with severe pneumonia, a RCT would now be possible. In the proposed study, we would identify under-5 children attending the outpatient department of the Radda Clinic and ICHSH with severe pneumonia and randomize them, in equal numbers, for management at the day-care centre (Radda Clinic) or hospital (ICHSH) subject to consent of respective parents/guardians. Children with very severe pneumonia, who needs hospitalization, would not be enrolled as they need hospital care and it would be unethical at this stage to enroll them in the proposed study. About 3000 children with a clinical diagnosis of pneumonia visit the clinic each year, and we estimate that about 200 of them will have severe pneumonia requiring hospitalization - the patient population of our study. We hope to enroll requisite 368 (184/site) children with severe pneumonia during 2-year study period.

ELIGIBILITY:
Inclusion Criteria:

* Age: 2 to 59 months
* Sex: Both boys and girls
* Severe pneumonia according to WHO criteria (Severe pneumonia is defined as cough or difficult breathing with lower chest wall in drawing with or without fast breathing which is defined as the respiratory rate ≥ 50 breaths per minute for children aged 2-11 months and ≥ 40 breaths per minute for children aged 12-59 months)
* Attend the Radda Clinic and ICHSH between 8:00 am to 4:00 pm (Sunday through Saturday)
* Written informed consent by respective parents/guardians

Exclusion Criteria:

* Very severe and non-severe pneumonia
* Nosocomial pneumonia
* History of taking antibiotics for pneumonia within 48 hour prior to enrollment
* Chronic illnesses like tuberculosis, cystic fibrosis
* Congenital deformities/anomalies e.g. Down's Syndrome, congenital heart disease
* Immunodeficiency
* Trauma/burn
* Bronchiolitis
* Bronchial asthma
* Lives far away from the Radda Clinic and ICHSH (outside 5 km radius from the respective study site)
* Parents/guardians not consenting for inclusion of their children in the study

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 368 (Estimated)
Dates: Start 2005-12; Primary Completion 2007-12 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Ashraf, MD, Principal Investigator — ICDDR,B: Centre for Health and Population Research
Locations (1):
- ICDDR,B, Dhaka, Bangladesh

REFERENCES:
- [Derived] Ashraf H, Alam NH, Chisti MJ, Salam MA, Ahmed T, Gyr N. Observational follow-up study following two cohorts of children with severe pneumonia after discharge from day care clinic/hospital in Dhaka, Bangladesh. BMJ Open. 2012 Jul 27;2(4):e000961. doi: 10.1136/bmjopen-2012-000961. Print 2012. PMID 22842561
- [Derived] Ashraf H, Mahmud R, Alam NH, Jahan SA, Kamal SM, Haque F, Salam MA, Gyr N. Randomized controlled trial of day care versus hospital care of severe pneumonia in Bangladesh. Pediatrics. 2010 Oct;126(4):e807-15. doi: 10.1542/peds.2009-3631. Epub 2010 Sep 20. PMID 20855397